CLINICAL TRIAL: NCT03379441
Title: A Randomized Phase II Study of Pembrolizumab (MK-3475) as Maintainance Therapy in Patients With Unresectable Stage III Non-small Cell Lung Cancer Treated With Definitive Chemo-radiotherapy
Brief Title: Pembrolizumab (MK-3475) as Maintainance in Treated Patients With Unresectable Stage III NSCLC
Acronym: MP-LALC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Prof. Silvia Novello, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-001252-22
Record Dates: First submitted 2017-11-23; First posted 2017-12-20 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Non Small Cell Lung Cancer Patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Pembrolizumab 200 mg Q3W IV infusion Day 1 of each 3 week cycle until:
  * PD,
  * unacceptable toxicity,
  * investigator choice,
  * patients IC withdrawal,
  * up to a maximum of 24 months (35 administrations) Experimental
  Interventions: Drug: Pembrolizumab Injectable Product
- Observation (No Intervention)

INTERVENTIONS:
Drug: Pembrolizumab Injectable Product — Pembrolizumab Injectable Product 200 mg Q3W Intravenous
  Arms: Experimental

SUMMARY:
Maintainance therapy in patients with unresectable stage III, NSCLC Stage IIIA-B, unresectable, NSCLC, treated with definitive Chemo-Radiotherapy

DETAILED DESCRIPTION:
This is an Italian multi-center randomized phase II trial (randomization 2:1) of intravenous (IV) MK-3475 (Pembrolizumab) versus observation as a maintenance therapy after chemo-radiotherapy (either concomitant or sequential, regardless of the type of chemotherapy used) in unresectable stage IIIA-IIIB non small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be > 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core, trucut biopsy or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the PI.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Section 8.14.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis, or has evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or Hepatitis C (e.g., HCV ribonucleic acid [RNA] qualitative is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
OS | up to 24 months per patient
  The primary objective is to evaluate if treatment with chemo-radiotherapy followed by Pembrolizumab (MK-3475) maintenance (up to 24 months) results in superior Overall Survival (OS) in stage IIIA-B, unresectable, NSCLC compared to chemo-radiotherapy (CT-RT) followed by observation

SECONDARY OUTCOMES:
PFS | up to 24 months per patient
  To evaluate Rate (%) of patients without disease progression at 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (14):
  - CRO Aviano, Aviano, Pordenone
  - AOU San Luigi- Department of Oncology, Orbassano, Turin
  - Istituto Tumori Giovanni Paolo II, Bari
  - Chieti Università degli Studi "G. D'Annunzio", Chieti
  - AOU Careggi, Florence
  - IRCCS AO San Martino, Genova
  - Azienda Ospedaliera Papardo, Messina
  - Istituto Clinico Humanitas, Milan
  - Ospedale San Raffaele, Milan
  - Policlinico Modena, Modena
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Policlinico Universitario Campus Biomedico, Roma
  - PO Centrale, Taranto
  - Policlinico Verona Borgo Roma, Verona